CLINICAL TRIAL: NCT07021040
Title: Analysis of Human Olfactory Biopsies
Brief Title: Olfactory Biopsies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00116591; 1R01DC021422-01A1 (NIH)
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Smell Loss; Smell Dysfunction
Keywords: act-seq; nasal biopsy; RNA-seq
MeSH Terms: conditions — Alzheimer Disease; Anosmia; Olfaction Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alzheimer's study (Other): Olfactory function will be assessed using the Smell Identification Test (SIT, Sensonics, Inc) or Sniffin' Sticks Test. Using topical intranasal decongestion/anesthetic (oxymetazoline/lidocaine), a cytology brush biopsy will be obtained from the olfactory cleft region of the nose in clinic exam room using a nasal endoscope.
  Interventions: Diagnostic Test: olfactory testing; Other: Odor stimulation; Procedure: Olfactory biopsy
- Act-seq study or Non-AD controls (Other): Olfactory function will be measured using established psychophysical testing via the Smell Identification Test or Sniffin' Sticks. Researchers will obtain biopsies from (1) normosmic subjects with or without odor stimulation, and (2) hyposmic subjects with history of upper respiratory infection (URI) as likely cause of the smell loss (such as COVID19) with or without odor stimulation.
  Interventions: Diagnostic Test: olfactory testing; Other: Odor stimulation; Procedure: Olfactory biopsy

INTERVENTIONS:
Diagnostic Test: olfactory testing — Patients will undergo smell testing, using the Smell Identification Test (Sensonics), a validated widely-used 40-item "scratch-and-sniff" style psychophysical test to determine olfactory function.
Other: Odor stimulation — subset of patients will be asked to sniff a specific odor for about an hour, using commercially available "odor pens" (Sniffin' Sticks or Sensonics). These odor pens are widely used for olfactory training therapy, a treatment designed to help people with some forms of smell loss; they are also used in psychophysical olfactory testing.
Procedure: Olfactory biopsy — Biopsy involves a simple cytology brush technique of the lining of the nose in a region called the olfactory cleft, using a nasal endoscope, and can be done in clinic or in the operating room at the time of a nasal surgery. Topical oxymetazoline and tetracaine spray is applied to the nasal cavity, a rigid nasal endoscopy (0-degree 4 mm endoscope, Karl Storz) is performed to visualize the olfactory cleft, and a small nasal cytology brush biopsy (Hobbs Medical)is performed by swabbing and rotating brush gently in the olfactory cleft. Cytology sample is placed into a buffer (Hibernate-E, Thermo Fisher)on ice for transport to the research lab.

SUMMARY:
This research study aims to investigate the function of the olfactory lining in the nasal cavity and its potential alterations in both healthy and diseased conditions. The olfactory lining is involved in the sense of smell.

The purpose of this study is to collect tissue from the nasal cavity.

DETAILED DESCRIPTION:
The purpose of this study is to analyze cell populations active in human olfactory tissue in health and disease. This is a prospective study. Healthy participants or participants with known disease processes that may impact olfaction, such as Alzheimer's, inflammatory conditions, aging, or post-viral smell loss, will be included. Olfaction will be measured using standard psychophysical testing. Biopsies of the olfactory lining in the nasal cavity may be obtained in the otolaryngology clinic or the operating room, if the patient is having an unrelated endoscopic nasal surgery, and may be obtained using a punch technique or a cytology brush. Before biopsies, some patients may be asked to sniff an odor substance (such as lavender, mint, citrus, or cloves) briefly, to stimulate olfactory cells. Biopsies will be processed for assays in the PI's lab, including histology, primary culture assays, flow cytometry assays, or transcriptomic profiling.

ELIGIBILITY:
Group 1: Alzheimer's study

Inclusion Criteria:

* Between the ages of 18 and 80
* Pre-clinical AD (this cohort consists of subjects who have normal cognitive testing and function, but have positive AD biomarkers);
* Symptomatic AD (a confirmed diagnosis of Alzheimer's or dementia who are capable of understanding and signing the consent document)

Exclusion Criteria:

* Advanced Alzheimer's/dementia
* Self-reported or known allergy to Afrin or Tetracain HCL (or related class of drugs)
* Active Rhinosinusitis symptoms
* Other known sinonasal disease history that would preclude biopsy (i.e prior sinus or skull base surgery directly impacting this anatomic region, sinonasal neoplasm in this anatomic region, olfactory cleft polyps)
* Parkinson's disease
* Unable or willing to complete the nasal endoscopy procedure.
* Unable to read or speak English
* Unable to provide legally effective consent

Group 2: Act-seq study or Non-AD controls

Inclusion Criteria:

* Age 18 years or older
* Patients being seen for rhinology or olfactory disorders
* Patients having unrelated endoscopic nasal surgery

Exclusion Criteria:

* Self-reported or known allergy to Afrin or Tetracain HCL (or related class of drugs)
* Unable or willing to complete the nasal endoscopy procedure
* Unable to read or speak English
* Unable to provide legally effective consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Transcription state changes in olfactory cells | study is planned for completion over 5 years
  Using single cell RNA-sequencing, olfactory epithelial cell populations will be analyzed for changes in coherent gene expression programs from subjects in different environmental conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Goldstein, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No